CLINICAL TRIAL: NCT05820347
Title: Validation of Inspiratory Muscle Pressure Estimation and Automated Detection of Asynchronies in Patients Under Assisted Mechanical Ventilation
Brief Title: Muscle Pressure Estimation With Artificial Intelligence During Mechanical Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Magnamed Tecnologia Medica S/A (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CAAE: 59353422.9.0000.0068
Record Dates: First submitted 2023-03-16; First posted 2023-04-19 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-03

CONDITIONS: Respiratory Failure
Keywords: mechanical ventilation; artificial intelligence
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Artificial Intelligence Estimation of Muscle Pressure during Mechanical Ventilation (Other): All included subjects will be monitored simultaneously with the esophageal balloon (gold standard) and with the artificial intelligence algorithm integrated in the mechanical ventilator. Electrical Impedance Tomography will be used to monitor ventilatory patterns during different degrees of spontaneous effort. First, a single intravenous bolus of neuromuscular blockade (succinylcholine 1mg/kg or rocuronium 1.2mg/kg) will be performed to measure respiratory system mechanics (compliance and resistance). In cases where rocuronium is used, a single dose of sugammadex 4mg/kg will be administered intravenously to reverse neuromuscular blockade after measuring compliance and resistance. After initiation of spontaneous breathing effort, pressure support will be titrated from 20 cmH2O to 2 cmH2O, in decremental steps during 20 minutes each. After completing titrating of pressure support, the esophageal balloon will be removed.
  Interventions: Device: Artificial Intelligence Estimation of Muscle Pressure during Mechanical Ventilation

INTERVENTIONS:
Device: Artificial Intelligence Estimation of Muscle Pressure during Mechanical Ventilation — Estimation of inspiratory muscle pressure by an artificial intelligence algorithm integrated in the mechanical ventilator (FlexiMag, Magnamed, Brazil).
  Other Names: Esophageal balloon measurements of Muscle Pressure; Transient Neuromuscular Blockade with Succinylcholine or Rocuronium to measure Respiratory Mechanics; Electrical Impedance Tomography Monitorization

SUMMARY:
The goal of this diagnostic study is to validate estimation of inspiratory muscle pressure by an artificial intelligence algorithm compared to the gold standard, the measure from an esophageal catheter balloon, in patients under assisted mechanical ventilation. The main questions it aims to answer are:

• Are inspiratory muscle pressure estimates from an artificial intelligence algorithm accurate when compared to the direct measure from an esophageal balloon?

Participants will be monitored with an esophageal balloon and with an artificial intelligence algorithm simultaneously, with inspiratory muscle pressure estimation during assisted mechanical ventilation with decremental levels of pressure support.

DETAILED DESCRIPTION:
This is a diagnostic study to validate estimation of inspiratory muscle pressure during assisted ventilation from an artificial intelligence algorithm integrated in a mechanical ventilator (FlexiMag, Magnamed, Brazil) compared to direct measure of muscle pressure from esophageal catheter balloon (gold standard). This is a novel non-invasive method to estimate inspiratory muscle pressure.

After obtaining informed consent, participants will be monitored simultaneously with the esophageal balloon and the artificial intelligence algorithm, with decremental levels of pressure support (20 to 2 cmH2O, in steps of 20 minutes). Esophageal balloon will be removed after completing the last pressure support step.

The investigators estimated a sample of 50 participants, considering 3 cmH2O as a clinically relevant discordance between methods and 10% of missing data. Concordance analysis and correlation analysis will be performed.

Procedures will follow a specific Standard Operating Procedures and participants inclusion data will be inserted in REDCap.

ELIGIBILITY:
Inclusion Criteria:

* Patients under assisted or assist-control mechanical ventilation

Exclusion Criteria:

* Contraindication to esophageal catheter insertion (esophageal cancer or bleeding, esophageal fistula, skull base fracture, uncontrolled coagulopathies)
* Contraindication to transient neuromuscular blockade
* Bronchopleural fistula (persistent air leak)
* Hemodynamic instability (norepinephrine > 1mcg/kg/min)
* Gestation
* Current sinus infection
* Refusal from patient's family of attending physician
* Palliative care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-08-26 (Actual); Primary Completion 2023-07-18 (Actual); Study Completion 2023-07-18 (Actual)

PRIMARY OUTCOMES:
Concordance between muscle pressure amplitude (in cmH2O) estimation by artificial intelligence and esophageal balloon | 4 hours
  Analysis of the bias and limits of agreement (Bland-Altman plot) between muscle pressure estimated amplitude in cmH2O from artificial intelligence and measured by esophageal balloon.
Correlation between muscle pressure amplitude estimation (in cmH2O) by artificial intelligence and esophageal balloon | 4 hours
  Correlation, reported as R-squared and a correlation plot, between amplitude in cmH2O of muscle pressure estimation by artificial intelligence and esophageal balloon.
Detection of initiation time and ending time of a spontaneous breathing cycle by artificial intelligence compared with esophageal balloon | 4 hours
  Time difference (in ms) between initiation of a spontaneous breathing cycle and ending of a spontaneous breathing cycle between artificial intelligence and esophageal balloon.

SECONDARY OUTCOMES:
Sensitivity and specificity of patient-ventilator asynchrony automated detection using the Artificial Intelligence Muscle Pressure estimator | 4 hours
  Number of patient-ventilator asynchronies detected using artificial intelligence compared with number of asynchronies detected by experts assessing airway pressure, flow and esophageal balloon waveforms.

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo LV Costa, MD, PhD, Principal Investigator — University of Sao Paulo; Marcelo BP Amato, MD, PhD, Study Chair — University of Sao Paulo
Locations (1):
- Heart Institute, University of São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amato MB, Barbas CS, Medeiros DM, Magaldi RB, Schettino GP, Lorenzi-Filho G, Kairalla RA, Deheinzelin D, Munoz C, Oliveira R, Takagaki TY, Carvalho CR. Effect of a protective-ventilation strategy on mortality in the acute respiratory distress syndrome. N Engl J Med. 1998 Feb 5;338(6):347-54. doi: 10.1056/NEJM199802053380602. PMID 9449727
- [Background] Acute Respiratory Distress Syndrome Network; Brower RG, Matthay MA, Morris A, Schoenfeld D, Thompson BT, Wheeler A. Ventilation with lower tidal volumes as compared with traditional tidal volumes for acute lung injury and the acute respiratory distress syndrome. N Engl J Med. 2000 May 4;342(18):1301-8. doi: 10.1056/NEJM200005043421801. PMID 10793162
- [Background] Loring SH, Malhotra A. Driving pressure and respiratory mechanics in ARDS. N Engl J Med. 2015 Feb 19;372(8):776-7. doi: 10.1056/NEJMe1414218. No abstract available. PMID 25693019
- [Background] Yoshida T, Torsani V, Gomes S, De Santis RR, Beraldo MA, Costa EL, Tucci MR, Zin WA, Kavanagh BP, Amato MB. Spontaneous effort causes occult pendelluft during mechanical ventilation. Am J Respir Crit Care Med. 2013 Dec 15;188(12):1420-7. doi: 10.1164/rccm.201303-0539OC. PMID 24199628
- [Background] Yoshida T, Roldan R, Beraldo MA, Torsani V, Gomes S, De Santis RR, Costa EL, Tucci MR, Lima RG, Kavanagh BP, Amato MB. Spontaneous Effort During Mechanical Ventilation: Maximal Injury With Less Positive End-Expiratory Pressure. Crit Care Med. 2016 Aug;44(8):e678-88. doi: 10.1097/CCM.0000000000001649. PMID 27002273
- [Background] Yoshida T, Amato MBP, Grieco DL, Chen L, Lima CAS, Roldan R, Morais CCA, Gomes S, Costa ELV, Cardoso PFG, Charbonney E, Richard JM, Brochard L, Kavanagh BP. Esophageal Manometry and Regional Transpulmonary Pressure in Lung Injury. Am J Respir Crit Care Med. 2018 Apr 15;197(8):1018-1026. doi: 10.1164/rccm.201709-1806OC. PMID 29323931
- [Background] Morais CCA, Koyama Y, Yoshida T, Plens GM, Gomes S, Lima CAS, Ramos OPS, Pereira SM, Kawaguchi N, Yamamoto H, Uchiyama A, Borges JB, Vidal Melo MF, Tucci MR, Amato MBP, Kavanagh BP, Costa ELV, Fujino Y. High Positive End-Expiratory Pressure Renders Spontaneous Effort Noninjurious. Am J Respir Crit Care Med. 2018 May 15;197(10):1285-1296. doi: 10.1164/rccm.201706-1244OC. PMID 29323536
- [Background] Sousa MLEA, Magrans R, Hayashi FK, Blanch L, Kacmarek RM, Ferreira JC. Clusters of Double Triggering Impact Clinical Outcomes: Insights From the EPIdemiology of Patient-Ventilator aSYNChrony (EPISYNC) Cohort Study. Crit Care Med. 2021 Sep 1;49(9):1460-1469. doi: 10.1097/CCM.0000000000005029. PMID 33883458
- [Background] Sousa MLA, Magrans R, Hayashi FK, Blanch L, Kacmarek RM, Ferreira JC. Predictors of asynchronies during assisted ventilation and its impact on clinical outcomes: The EPISYNC cohort study. J Crit Care. 2020 Jun;57:30-35. doi: 10.1016/j.jcrc.2020.01.023. Epub 2020 Jan 21. PMID 32032901
- [Background] Blanch L, Villagra A, Sales B, Montanya J, Lucangelo U, Lujan M, Garcia-Esquirol O, Chacon E, Estruga A, Oliva JC, Hernandez-Abadia A, Albaiceta GM, Fernandez-Mondejar E, Fernandez R, Lopez-Aguilar J, Villar J, Murias G, Kacmarek RM. Asynchronies during mechanical ventilation are associated with mortality. Intensive Care Med. 2015 Apr;41(4):633-41. doi: 10.1007/s00134-015-3692-6. Epub 2015 Feb 19. PMID 25693449
- [Background] LeCun Y, Bengio Y, Hinton G. Deep learning. Nature. 2015 May 28;521(7553):436-44. doi: 10.1038/nature14539. PMID 26017442
- [Background] Pletsch-Assuncao R, Caleffi Pereira M, Ferreira JG, Cardenas LZ, de Albuquerque ALP, de Carvalho CRR, Caruso P. Accuracy of Invasive and Noninvasive Parameters for Diagnosing Ventilatory Overassistance During Pressure Support Ventilation. Crit Care Med. 2018 Mar;46(3):411-417. doi: 10.1097/CCM.0000000000002871. PMID 29189344
- [Background] Baydur A, Behrakis PK, Zin WA, Jaeger M, Milic-Emili J. A simple method for assessing the validity of the esophageal balloon technique. Am Rev Respir Dis. 1982 Nov;126(5):788-91. doi: 10.1164/arrd.1982.126.5.788. PMID 7149443
- [Background] Liao JJ. Sample size calculation for an agreement study. Pharm Stat. 2010 Apr-Jun;9(2):125-32. doi: 10.1002/pst.382. PMID 19507134
- [Background] Motta APG, Rigobello MCG, Silveira RCCP, Gimenes FRE. Nasogastric/nasoenteric tube-related adverse events: an integrative review. Rev Lat Am Enfermagem. 2021 Jan 8;29:e3400. doi: 10.1590/1518-8345.3355.3400. eCollection 2021. PMID 33439952